CLINICAL TRIAL: NCT00486213
Title: Randomized Double-Blind Placebo-Controlled Trial of Pyridoxine for Prevention of Capecitabine-Induced Hand-Foot Syndrome (HFS)
Brief Title: Pyridoxine in Preventing Hand-Foot Syndrome Caused by Capecitabine in Patients With Cancer
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Slow accrual
Sponsor: National Cancer Centre, Singapore (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: CDR0000551757; SINGAPORE-06-22-OTH
Record Dates: First submitted 2007-06-13; First posted 2007-06-14 (Estimated); Last update posted 2015-09-24 (Estimated); Status verified 2015-09

CONDITIONS: Dermatologic Complications; Palmar-plantar Erythrodysesthesia; Unspecified Adult Solid Tumor, Protocol Specific
Keywords: dermatologic complications; chemotherapeutic agent toxicity; palmar-plantar erythrodysesthesia; unspecified adult solid tumor, protocol specific
MeSH Terms: conditions — Hand-Foot Syndrome | interventions — Pyridoxine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Pyridoxine hydrochloride (Active Comparator): Pyridoxine (200mg) or placebo once daily orally for 21 days out of each treatment cycle
  Interventions: Dietary Supplement: pyridoxine hydrochloride
- Placebo (Placebo Comparator): Pyridoxine (200mg) or placebo once daily orally for 21 days out of each treatment cycle
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: pyridoxine hydrochloride — Pyridoxine (200mg) or placebo once daily orally for 21 days out of each treatment cycle
  Arms: Pyridoxine hydrochloride
Other: Placebo
  Arms: Placebo

SUMMARY:
RATIONALE: Pyridoxine may help prevent hand-foot syndrome caused by capecitabine in patients with cancer. It is not yet known whether pyridoxine is more effective than a placebo in preventing hand-foot syndrome in patients with cancer.

PURPOSE: This randomized phase III trial is studying pyridoxine to see how well it works compared with a placebo in preventing hand-foot syndrome caused by capecitabine in patients with cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Compare the incidence of capecitabine-induced palmar-plantar erythrodysesthesia (hand-foot syndrome [HFS]) ≥ grade 2 in patients with cancer treated with pyridoxine hydrochloride vs placebo.

Secondary

* Compare the time to onset of HFS ≥ grade 2 in patients treated with these regimens.
* Compare the quality of life changes in patients treated with these regimens.
* Identify factors predicting toxicity from capecitabine chemotherapy.

OUTLINE: This is a randomized, double-blind, placebo-controlled study. Patients are stratified according to gender and treatment setting (adjuvant/neoadjuvant vs palliative setting). Patients are randomized to 1 of 2 treatment arms.

* Arm I: Beginning concurrently with planned capecitabine treatment, patients receive oral pyridoxine hydrochloride once daily on days 1-21.
* Arm II: Beginning concurrently with planned capecitabine treatment, patients receive oral placebo once daily on days 1-21.

In both arms, treatment repeats every 21 days for up to 8 courses (until discontinuation of capecitabine treatment).

Quality of life is assessed at baseline, at the beginning of courses 2, 4, 6, and 8, and at the end of the study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of cancer
* Must be receiving single-agent capecitabine either in the adjuvant/neoadjuvant or palliative setting at a dose of ≥ 1000 mg/m² twice daily on days 1-14 (given in 3-week courses)

PATIENT CHARACTERISTICS:

* Life expectancy > 12 weeks
* No preexisting neuropathy
* No known allergy to pyridoxine hydrochloride and its incipients
* No other dermatologic condition that, in the opinion of the physician, may affect the hands or feet or may complicate evaluation during study treatment

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No prior capecitabine
* Concurrent radiotherapy, steroids, and/or biological therapy (e.g., trastuzumab [Herceptin®] or bevacizumab) allowed provided they do not cause hand-foot syndrome (HFS)
* No other concurrent drugs (e.g., docetaxel or doxorubicin hydrochloride liposome) that can cause HFS
* No concurrent drugs (e.g., oxaliplatin or taxanes) that can cause neuropathy
* No concurrent pyridoxine hydrochloride-containing preparations (e.g., multivitamins or vitamin B complex)
* No concurrent over-the-counter products that contain urea or lactic acid
* No concurrent drugs reported to have drug interactions with pyridoxine hydrochloride (e.g., cycloserine; hydralazine; immunosuppressants; isoniazid; levodopa; estrogen or estrogen-containing contraceptives; penicillamine; phenobarbitone; phenytoin; or pyrazinamide)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Actual)
Dates: Start 2007-06; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
First incidence of hand-foot syndrome (HFS) ≥ grade 2 according to NCI CTCAE vs 3.0 | up to 8 cycles

SECONDARY OUTCOMES:
Time to the onset of HFS ≥ grade 2 | days to weeks
Quality of life as measured by EuroQOL (EQ-5D) questionnaire | QOL assessment at baseline, at beginning of cycles 2, 4, 6, 8 and at the end of the study.

CONTACTS AND LOCATIONS:
Overall Officials: Yoon-Sim Yap, FRACP, MBBS, Principal Investigator — National Cancer Centre, Singapore
Locations (1):
- National Cancer Centre - Singapore, Singapore, Singapore

REFERENCES:
- [Derived] Yap YS, Kwok LL, Syn N, Chay WY, Chia JWK, Tham CK, Wong NS, Lo SK, Dent RA, Tan S, Mok ZY, Koh KX, Toh HC, Koo WH, Loh M, Ng RCH, Choo SP, Soong RCT. Predictors of Hand-Foot Syndrome and Pyridoxine for Prevention of Capecitabine-Induced Hand-Foot Syndrome: A Randomized Clinical Trial. JAMA Oncol. 2017 Nov 1;3(11):1538-1545. doi: 10.1001/jamaoncol.2017.1269. PMID 28715540